CLINICAL TRIAL: NCT07229287
Title: Effects of Kinetic Control Training on Pain, Postural Stability, Gait and Endurance in Patients With Chronic Sacroiliac Joint Dysfunction
Brief Title: Kinetic Control Exercises to Reduce Pain and Improve Balance, Walking, and Stamina in Sacroiliac Joint Issues
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Manum Tahir, Principal Investigator (Clinical Musculoskeletal Physiotherapist, Faculty of Rehabilitation Sciences), Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FORS/25/026; UBAS/ERB/FORS/25/026 (Other: Lahore University of Biological and Applied Sciences)
Record Dates: First submitted 2025-10-01; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Low back pain; Sacroiliac joint dysfunction; Pelvic girdle pain
MeSH Terms: conditions — Low Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- movement retraining with the concept of kinetic control (Experimental): The interventional group receives Kinetic control training, which target two muscle groups mainly abdominals and glutes along with usual treatment
  Interventions: Other: movement retraining/ kinetic control; Other: Routine Physical therapy
- Routine Physical Therapy Intervention for sacroilliac joint dysfunction (Active Comparator): Routine physical therapy intervention includes, hot pack for 15 mins and exercise therapy for 25 mins, including sacroiliac joint self-mobilization, piriformis, gluteus medius, minimums, and maximus stretches, isometric hip exercises, knee-to-shoulder stretch, quadriceps and hamstring stretches, back-bridge.
  Interventions: Other: Routine Physical therapy

INTERVENTIONS:
Other: movement retraining/ kinetic control — this intervention is for experimental group. Kinetic control is grounded in the principles of motor control training and movement retraining. In this study, this intervention primarily focuses on activating and strengthening two key muscle groups: the abdominals and obliques, along with the gluteal muscles.
  Arms: movement retraining with the concept of kinetic control
Other: Routine Physical therapy — Routine physical therapy intervention will be given to the patient which includes, hot pack for 15 mins and exercise therapy for 25 mins, involving floor sessions including sacroiliac joint self-mobilization, piriformis, gluteus medius, minimums, and maximus stretches, leg pressing inward/outward, knee-to-shoulder stretch, quadriceps and hamstring stretches, standard and one-leg elevated

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the Kinetic control on pain, endurance, Gait and postural stability in patients suffering from chronic sacroiliac joint dysfunction.

The main question it aims to answer is:

* Does kinetic control training work on pain in SIJ dysfunction?
* Does kinetic control therapy work on functional outcomes, including gait metrics, postural sway, and lumbar endurance?

The treatment arm will receive the Kinetic control training, and the comparison arm will undergo standard physical therapy care. Participants will be asked to perform movement control exercises based on the principle of kinetic control training core muscles and hip muscles after routine physical therapy. The participants in the control/comparison group will only receive routine physical therapy that includes a heating pad, TENS, joint mobilizations, and stretching and strengthening exercises.

DETAILED DESCRIPTION:
The sacroiliac joint connects the lower part of the spine (sacrum) to the pelvic bones (ilium) and helps transfer body weight between the upper body and legs. It plays an important role in providing stability while allowing limited movement during walking or bending.

Sacroiliac joint dysfunction (SIJD) occurs when the joint becomes inflamed, stiff, or moves abnormally. This may cause pain in the lower back, buttocks, or thighs, sometimes spreading to the groin or legs. People with SIJD often experience difficulty standing for long periods, walking, or bending. The condition is commonly mistaken for lumbar spine or hip problems because of overlapping symptoms. Research shows that 15-30% of people with long-term lower back pain may actually have SIJ dysfunction, but many cases go undiagnosed due to the absence of a single definitive test.

Kinetic control is a movement-based physiotherapy method that focuses on retraining how muscles coordinate to stabilize and move joints. It aims to correct poor movement control, improve muscle endurance, and restore healthy patterns of motion, particularly in the core and hip muscles. By improving control and alignment, kinetic control training may reduce pain and enhance posture, walking ability, and overall function.

In this 8-week randomized controlled trial, participants with chronic SIJ dysfunction will be assigned to one of two groups. The intervention group will receive kinetic control-based exercises in addition to routine physiotherapy, while the control group will receive standard physiotherapy treatments such as heat therapy, TENS, joint mobilizations, stretching, and strengthening exercises.

Assessments will be conducted at the beginning, after 4 weeks, and after 8 weeks, measuring pain, balance, gait, and lumbar muscle endurance using validated tools. The study aims to determine whether kinetic control provides greater improvements in pain relief, postural control, walking performance, and endurance compared to routine care in individuals with chronic sacroiliac joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of sacroiliac joint dysfunction lasting more than 2 months
* Male and female participants aged 20-60 years
* Positive lumbopelvic motor control tests
* Pain intensity of ≥4 on a 0-10 Numeric pain rating scale (NPRS)
* Positive results in three or more of the following provocative tests: FABER test, Distraction test, Thigh Thrust test, Gaenslen test, or Sacral Thrust test
* Diagnosis consistent with International Association for the Study of Pain (IASP) criteria, indicating pain localized to the sacroiliac joint region (hips/groins or radiating to the lower extremity)

Exclusion Criteria:

* History of malignancy
* Neurological disease affecting the central nervous system (e.g., multiple sclerosis, dementia)
* Rheumatic disease (e.g., fibromyalgia, ankylosing spondylitis, rheumatoid arthritis)
* Disc herniation or lumbar radiculopathy due to systemic disease
* Spinal surgery within the last 12 months
* Pregnancy
* Signs or symptoms of lumbar nerve root pathology identified during neurological examination

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Intensity Measured by the Numeric Pain Rating Scale (NPRS) at 4 and 8 Weeks | From enrollment to 4 weeks, then at the end of 8 weeks
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), where participants rate their pain on a scale ranging from 0 to 10 units (Unit of Measure: score on a 0-10 scale). A score of 0 represents no pain, while 10 indicates the worst imaginable pain. Pain severity will be categorized as mild (1-3), moderate (4-6), and severe (7-10) A decrease in NPRS score from baseline will indicate an improvement in pain intensity, whereas higher scores will reflect greater pain severity.
Change from Baseline in Postural Stability Measured by the Single-Leg Stance Test at 4 and 8 Weeks | From enrollment to 4 weeks, then at the end of 8 weeks
  Postural stability will be evaluated using the Single-Leg Stance Test (SLST), which measures the participant's ability to maintain balance on one leg without support. The duration of balance maintenance will be recorded in seconds (unit of measure: seconds [s]). Each participant will perform three trials, and the mean value of the three measurements will be used for analysis to ensure accuracy and consistency. Higher mean values indicate better postural control and balance, whereas lower values reflect reduced stability or impaired balance performance.
Change from Baseline in Lumbar Muscle Endurance Measured by Pressure Biofeedback Unit at 4 and 8 Weeks | From enrollment to 4 weeks, and then at the end of 8 weeks
  Lumbar muscle endurance will be assessed using a Pressure Biofeedback Unit (PBU) to evaluate the ability of the deep core stabilizing muscles to maintain a target pressure during a sustained contraction. The duration (in seconds) that participants can maintain the target pressure of 40-60 mmhg without deviation will be recorded (unit of measure: seconds [s]). Each participant will perform three trials, and the mean value of the three measurements will be used for analysis to enhance reliability.
  Higher mean endurance times will indicate better lumbar muscle endurance and motor control, while lower times will reflect fatigue or weakness of the stabilizing muscles.
Change from Baseline in Gait Parameters Measured by Kinovea Motion Analysis Software at 4 and 8 Weeks | From enrollment to 4 weeks, then at the end of 8 weeks
  Gait performance will be analyzed using Kinovea motion analysis software, which will capture and calculate spatiotemporal gait parameters. The parameters to be measured include step length (centimeters [cm]), stride length (centimeters [cm]), cadence (steps per minute [steps/min]), and walking speed (meters per second [m/s]) (Unit of Measure: cm, steps/min, m/s). Each participant will perform three walking trials at a self-selected comfortable speed, and the mean value of the three trials will be used for analysis to ensure measurement reliability.
  Increases in step length, stride length, cadence, and walking speed will indicate improved gait performance and functional mobility, whereas decreases in these parameters will reflect reduced gait efficiency or impaired locomotor control.

SECONDARY OUTCOMES:
Change from Baseline in Functional Disability Measured by the Modified Oswestry Disability Index (MODI) at 4 and 8 Weeks. | From enrollment to 4 weeks, then at the end of 8 weeks
  Functional disability will be assessed using the Modified Oswestry Disability Index (MODI), a validated questionnaire designed to measure limitations in daily living activities caused by low back or sacroiliac joint pain. The MODI consists of 10 sections, each scored from 0 to 5, with the total score converted into a percentage representing the level of disability (Unit of Measure: percentage [%]). The overall score ranges from 0% to 100%, where 0% indicates no disability and 100% indicates maximum disability. Disability levels are categorized as minimal (0-20%), moderate (21-40%), severe (41-60%), crippled (61-80%), and bed-bound (81-100%).
  A decrease in MODI percentage score will indicate improvement in functional ability and reduction in disability, while higher scores will reflect greater functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Manum Tahir, Study Director — Lahore University of Biological and Applied Sciences
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan